CLINICAL TRIAL: NCT00045812
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled, Study to Evaluate SCH-58235 in Homozygous Sitosterolemia
Brief Title: SCH-58235 (Ezetimibe) to Treat Homozygous Sitosterolemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 010115; 01-H-0115
Record Dates: First submitted 2002-09-10; First posted 2002-09-11 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2004-04

CONDITIONS: Lipoidosis
Keywords: Cholesterol; Sitosterol; Atherosclerosis; Intestine; Absorption; Homozygous Sitosterolemia; Sterol Metabolism
MeSH Terms: conditions — Lipidoses; Atherosclerosis | interventions — Ezetimibe

INTERVENTIONS:
Drug: SCH-58235

SUMMARY:
This study will test the safety and effectiveness of SCH-58235 (Ezetimibe) in lowering sitosterol, plant sterol and cholesterol blood levels in patients with homozygous sitosterolemia when added to the patients' current treatment regimen. Homozygous sitosterolemia is an inherited disorder of sterol metabolism in which an excess of many plant sterols, including sitosterol, is absorbed and not enough excreted. (Sterols are substances used to form hormones, vitamins and membranes found in animal and plant lipids.). Patients can develop atherosclerosis with coronary heart disease as early as childhood, as well as other problems including arthritis, arthralgia, and tendon xanthomas (lipid deposits). Current sitosterolemia treatments may include a low sterol diet, medications, intestinal surgery, or a combination of these. Ezetimibe is a member of a new class of drugs called "specific cholesterol absorption inhibitors" that may lower cholesterol, sitosterol and other plant sterol blood levels.

Patients with homozygous sitosterolemia 10 years of age and older may be eligible for this study. Participants will have a medical history and physical examination and will be randomly assigned to one of two treatment groups. One group, which will include about 80 percent of all study participants, will take 10 mg of Ezetimibe a day, and the second group (20 percent of participants) will take a placebo (an inactive look-a-like pill).

Patients will have 7 clinic visits during the 12-week study, when some or all of the following procedures and tests will be done:

* Measurement of vital signs (heart rate, blood pressure, breathing rate and temperature)
* Dietary maintenance - interview about how well that patient is adhering to the diet
* Medication review - interview about other medications the patient is taking
* Blood draw for tests
* Urine sample for tests
* Pregnancy test for women of childbearing potential
* Electrocardiogram (ECG) to measure the electrical activity of the heart
* Blood draw to determine sitosterol, other plant sterol levels, and lipid levels (cholesterol and other blood lipid concentrations)
* Xanthoma measurement (with a ruler and X-ray of the foot)

DETAILED DESCRIPTION:
Homozygous sitosterolemia is an autosomally inherited recessive disorder of sterol metabolism. Patients with homozygous sitosterolemia can present with accelerated atherosclerosis with initial CHD events occurring in childhood. In addition, these patients can have tendon xanthomas, hemolytic episodes, as well as arthritis and arthralgias. Plasma levels of sitosterol and other dietary sterols are markedly elevated in homozygous sitosterolemic patients, and are diagnostic of this disorder. A low sterol diet provides only limited reduction in sitosterol levels and currently available medical treatments, such as bile salt binding resins, are usually insufficiently effective or poorly tolerated.

SCH-58235 is a member of a new class of therapeutic agents, specific cholesterol absorption inhibitors, being developed to treat hypercholesterolemia. Preclinical animal studies and clinical studies in humans have demonstrated significant reductions in serum cholesterol levels with SCH-58235 treatment. In the current study, the efficacy and safety of SCH-58235 will be studied in patients with homozygous sitosterolemia, an inherited condition in which a wide range of plant sterols, including sitosterol, are excessively absorbed and inadequately excreted, leading to dramatic increases in tissue deposition. SCH-58235 may lower sitosterol levels by directly inhibiting sitosterol absorption (since plant sterols and cholesterol are structurally similar sterols) and/or by inhibiting cholesterol absorption and indirectly by increasing hepatic uptake of plasma LDL with increased cholesterol and sitosterol excretion. These mechanisms of action could lead to reductions in both plant sterol and LDL cholesterol levels in these patients, thereby providing important clinical benefits. The current study will determine if SCH-58235 will be safe and well tolerated and provide significant reductions in plant sterols (plasma sitosterol and campesterol) and low-density lipoprotein-cholesterol (LDL-C) concentrations in patients with homozygous sitosterolemia.

This is a multicenter, randomized, double-blind, placebo-controlled study lasting 12 weeks. Patients with a diagnosis of homozygous sitosterolemia who have an elevated plasma sitosterol level on their current regimen will be studied. Patients will be eligible to enroll in the study whether their current regimen is medication(s), surgical (prior ileal bypass), apheresis, a combination of treatments, or no active regimen. The primary objective of this study is to evaluate the efficacy and safety of 10 mg/day of SCH-58235 in patients with homozygous sitosterolemia who continue to have an elevated plasma sitosterol level.

ELIGIBILITY:
INCLUSION/EXCLUSION CRITERIA

Male or female, age greater than or equal to 10 years are eligible.

Patients must have a diagnosis of homozygous sitosterolemia with an elevated plasma sitosterol level (greater than 5 mg/dL at screening visit) on their current regimen.

All women of childbearing potential must be practicing an effective method of contraception.

All women of childbearing potential must have a negative urine pregnancy test within 72 hours prior to the start of the study medication.

Patients must not have any condition which, in the opinion of the investigator, would be likely to render the patient unable to complete the study or for which study participation would produce significant risk or not be in the best interests of the patient.

Individual with poor mental function, drug or substance abuse, or individuals with unstable psychiatric illness, which, in the opinion of the investigator, may interfere with optimal participation in the study will be excluded.

Women must not be pregnant or lactating.

Patients must not have had treatment with any other investigational drug within 30 days prior to visit 1.

Patients can not newly diagnosed or untreated person who has not been given an opportunity to consider treatment with standard of care and an opportunity to decline such treatment.

Patients must not have congestive heart failure NYHA class III or IV.

Patients must not have uncontrolled cardiac arrhythmias.

Patients must not have had a myocardial infarction, coronary bypass surgery or angioplasty within 6 months of the screening visit (Visit 1).

Patients must not have unstable angina pectoris or unstable or severe peripheral vascular disease.

Patients must not have uncontrolled diabetes mellitus (Hb(A1c) greater than 10%). Patients with diabetes mellitus should be on a stable antihyperglycemic regimen for at least 4 weeks prior to the screening visit (Visit 1).

Patients must not have uncontrolled endocrine or metabolic disease known to influence serum lipids or lipoproteins. Clinically euthyroid patients on stable replacement doses of thyroid hormone (on the same dose for at least 4 weeks prior to study entry and with TSH equal to 10 IU/mL) are eligible for enrollment.

Patients must not have uncontrolled hypertension (systolic BP greater than 200 mm Hg and/or diastolic BP greater than 110 mm Hg).

Patients must not have creatinine greater than 2.0 mg/dL at the screening visit (Visit 1), or active renal disease with significant proteinuria (greater than 1 albumin/mg creatinine).

Patients must not have active acute or chronic hepatobiliary disease; AST or ALT greater than 5 times the upper limit of normal of the reference laboratory at the screening visit (Visit 1).

Patients must not have disorders of the hematologic, digestive (including malabsorptive disorders), or central nervous system including cerebrovascular disease and degenerative diseases that would limit study evaluation or participation.

Patients must not be HIV positive.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 5
Dates: Start 2001-03; Study Completion 2004-04

CONTACTS AND LOCATIONS:
Locations (1):
- National Heart, Lung and Blood Institute (NHLBI), Bethesda, Maryland, United States

REFERENCES:
- [Background] Salen G, Shefer S, Nguyen L, Ness GC, Tint GS, Shore V. Sitosterolemia. J Lipid Res. 1992 Jul;33(7):945-55. PMID 1431587
- [Background] Bhattacharyya AK, Connor WE, Lin DS, McMurry MM, Shulman RS. Sluggish sitosterol turnover and hepatic failure to excrete sitosterol into bile cause expansion of body pool of sitosterol in patients with sitosterolemia and xanthomatosis. Arterioscler Thromb. 1991 Sep-Oct;11(5):1287-94. doi: 10.1161/01.atv.11.5.1287. PMID 1911714